CLINICAL TRIAL: NCT04580420
Title: A Phase 2 Open-Label Study to Evaluate the Safety and Efficacy of DCR-PHXC in Patients With Primary Hyperoxaluria Type 1 and Severe Renal Impairment, With or Without Dialysis
Brief Title: Safety & Efficacy of DCR-PHXC in Patients With PH1 and ESRD
Acronym: PHYOX7
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DCR-PHXC-204
Record Dates: First submitted 2020-09-24; First posted 2020-10-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Hyperoxaluria Type 1; End Stage Renal Disease
Keywords: PH1; ESRD
MeSH Terms: conditions — Primary hyperoxaluria type 1; Kidney Failure, Chronic | interventions — nedosiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label DCR-PHXC (Experimental): Open-Label monthly subcutaneous injection of DCR-PHXC based on age and weight.
  Interventions: Drug: DCR-PHXC

INTERVENTIONS:
Drug: DCR-PHXC — Monthly dosing throughout study period
  Other Names: Nedosiran

SUMMARY:
The aim of this study is to evaluate DCR-PHXC in participants with PH1 and severe renal impairment, with or without dialysis.

DETAILED DESCRIPTION:
The DCR-PHXC-204 study is listed under study number NN7022-8398 in Novo Nordisk systems.

This is an open-label, repeat-dose, Phase 2 study of DCR-PHXC in participants with PH1 and severe renal impairment, with or without dialysis. Following the up-to-35- day screening period, participants will return to the clinic for monthly dosing visits through Day 180. Participants successfully completing the Day 180 visit will continue on to an extended follow-up period and receive open-label DCR-PHXC for an additional 5 years, or until DCR-PHXC is commercially available, whichever comes first. As participants in this extended treatment period will return to the clinic only every 3 months, participants and/or their caregivers may be trained in the at-home administration of DCR-PHXC or home health nurses may assist with administration of DCR -PHXC.

The total duration of the study is approximately 5 years from first participant, first visit, to last participant, last Day 180 visit, with up to an additional 5 years of extended follow-up.

ELIGIBILITY:
Note: Currently, the DCR-PHXC-204 study is only enrolling potential participants under 6 years of age.

Inclusion Criteria:

1. Four age groups of participants will be enrolled:

   1. adults and adolescents (aged ≥ 12 years)
   2. children 6 to 11 years of age
   3. children 2 to 5 years of age
   4. infants and newborns from birth to < 2 years of age
2. . Documented diagnosis of PH1, confirmed by genotyping
3. Estimated GFR at Screening <30mL/min normalized to 1.73m^2 BSA
4. Mean of 2 Plasma Oxalate >20μmol/L during screening
5. For participants receiving hemodialysis or peritoneal dialysis total duration of hemodialysis or peritoneal dialysis must be less than 24 months and hemodialysis or peritoneal dialysis regimen must have been stable for at least 2 weeks prior to Screening.
6. Male or Female

   1. Male participants:

      * A male participant with a female partner of childbearing potential must agree to use contraception during the treatment period and for at least 12 weeks after the last dose of study intervention and refrain from donating sperm during this period.
   2. Female participants:

      * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

      Not a woman of childbearing potential (WOCBP).
      * OR
      * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 12 weeks after the last dose of study intervention and agrees to refrain from harvesting/freezing eggs during this period.
   3. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
7. Participant (and/or participant's parent or legal guardian if participant is a minor [defined as patient <18 years of age, or younger than the age of majority according to local regulations]) is capable of giving signed informed consent, which includes compliance with the requirement and restrictions listed in the informed consent form (ICF) and in the protocol.

   1. Adolescents (12 to < 18 years of age, or older than 12 years but younger than the age of majority according to local regulations) must be able to provide written assent for participation.
   2. For children younger than 12 years of age, assent will be based on local regulations
8. Affiliated with or is a beneficiary of a health insurance system (if applicable per national regulations)

Exclusion Criteria:

1. Prior hepatic transplantation; or scheduled transplantation within 6 months of Day 1. Prior renal transplantation is allowed.
2. Documented evidence of clinical manifestations of severe systemic oxalosis (including preexisting retinal, heart, or skin calcifications, or history of severe bone pain, pathological fractures, or bone deformations)
3. Presence of any condition or comorbidities that would interfere with study compliance or data interpretation or potentially impact patient safety including, but not restricted to:

   1. Severe intercurrent illness
   2. Known causes of active liver disease/injury (e.g., alcoholic liver disease, nonalcoholic fatty liver disease/steatohepatitis)
   3. Non-PH related conditions contributing to renal insufficiency
   4. Physician concerns about intake of drugs of abuse or excessive alcohol intake, or history of excessive alcohol intake in the 2 years prior to enrollment (defined as ≥ 21 units of alcohol per week in men and ≥ 14 units of alcohol per week in women; where a "unit" of alcohol is equivalent to a 12-ounce beer, 4-ounce glass of wine, or 1ounce shot of hard liquor)
4. Use of an RNAi drug, other DCR-PHXC, within the last 6 months
5. History of one or more of the following reactions to an oligonucleotide-based therapy:

   1. Severe thrombocytopenia (platelet count ≤ 100,000/µL)
   2. Hepatotoxicity, defined as alanine transaminase (ALT) or aspartate transaminase (AST) > 3 times the upper limit of normal (ULN) and total bilirubin > 2 × ULN or international normalized ratio (INR) >1.5
   3. Severe flu-like symptoms leading to discontinuation of therapy
   4. Localized skin reaction from the injection (graded severe) leading to discontinuation of therapy
   5. Coagulopathy/clinically significant prolongation of clotting time
6. Participation in any clinical study in which they received an investigational medicinal product (IMP) other than DCR-PHXC within 4 months before Screening.
7. Liver function test abnormalities: ALT and/or AST >1.5 × ULN for age and gender
8. Positive anti-double-stranded deoxyribonucleic acid (anti-dsDNA) antibody test at Screening
9. Known hypersensitivity to DCR-PHXC or any of its ingredients
10. Inability or unwillingness to comply with the specified study procedures, including the lifestyle considerations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2031-12-30 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of Events | 180 days
  To assess the efficacy of DCR-PHXC in lowering Pox in participants with PH1 and severe renal impairment, with or without hemodialysis or peritoneal dialysis.
Safety: Incidence of Events | 180 days
  Characterize the safety of DCR-PHXC in participants with PH1 and severe renal impairment, with or without dialysis.

SECONDARY OUTCOMES:
Change from Baseline in Plasma Oxalate Concentration | 180 Days
  To evaluate the effect of DCR-PHXC on Plasma Oxalate concentration from Baseline to day 180
To characterize the PK of DCR PHXC in patients with PH by observing secondary parameters of the area under the curve. | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including secondary parameters of area under the curve (AUC)
To characterize the PK of DCR PHXC in patients with PH by observing maximum observed concentration (Cmax). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including maximum observed concentration (Cmax)
To characterize the PK of DCR PHXC in patients with PH by observing minimum concentration (Cmin). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including minimum observed concentration (Cmin)
To characterize the PK of DCR PHXC in patients with PH by observing maximum concentration (Tmax). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including time to maximum concentration (Tmax)
To characterize the PK of DCR PHXC in patients with PH by observing terminal elimination half-life (t1/2). | 180 days
  Population and individual pharmacokinetic (PK) parameters for DCR PHXC, including terminal elimination half-life (t1/2)
Change in Frequency of Dialysis | 180 days
  Change from Baseline in the frequency of dialysis over 180 days
Change in Duration of Dialysis | 180 days
  Change from Baseline in the duration of dialysis over 180 days

OTHER OUTCOMES:
Change from Baseline in the Short Form (36) Health Survey (SF-36®) in adults | 180 days
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The SF 36 is a set of generic, coherent, and easily administered quality-of-life measures that taps 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. The 36 items are identical to the MOS SF 36 described in Ware and Sherbourne (1992). Participants respond to each item on a categorical scale. Categorical answers are transformed to a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. All items are scored so that a high score defines a more favorable health state
Change from Baseline in the EQ-5D-5L™ in adults | 180 days
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The EQ-5D-5L consists of the EQ 5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The digits for the 5 dimensions can be combined into a 5-digit number that describes the participant's health state.
  The EQ VAS records the participant's self-rated health on a 20-cm vertical VAS, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine.' Participants are asked to place an "X" on the line that represents their health on that day.
Change from Baseline in the Pediatric Quality of Life Inventory (PedsQL™) in children | 180 days
  To evaluate the effect of DCR-PHXC on Quality of Life (QoL) assessments in patients with PH.
  The 23-item PedsQL is comprised of 5 items in the Emotional, Social, and School Functioning dimensions (Psychosocial Health) and 8 items in the Physical Functioning (Physical Health) dimension. Items are reverse-scored on a 0 to 4 Likert scale and linearly transformed to a 0 to 100 scale, so that higher scores indicate better functioning and HRQOL. Scale Scores are the sum of the items in each dimension, divided by the number of items answered.
Changes from Baseline number of kidney stones | 180 days
  Evaluate the effect of DCR-PHXC on stone burden in participants with PH1 and severe renal impairment through Kidney Ultrasound
Changes from Baseline size of kidney stones | 180 days
  Evaluate the effect of DCR-PHXC on stone burden in participants with PH1 and severe renal impairment through Kidney Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (16):
- United States (4):
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
- France (2):
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Paris
- Germany (2):
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Heidelberg
- Clinical Trial Site, Roma, Italy
- Clinical Trial Site, Beirut, Lebanon
- Clinical Trial Site, Casablanca, Morocco
- Clinical Trial Site, Oradea, Romania
- Spain (2):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Santa Cruz de Tenerife
- Clinical Trial Site, Dubai, United Arab Emirates
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox JH, Boily MO, Caron A, Sheng T, Wu J, Ding J, Gaudreault S, Chong O, Surendradoss J, Gomez R, Lester J, Dumais V, Li X, Gumpena R, Hall MD, Waterson AG, Stott G, Flint AJ, Moore WJ, Lowther WT, Knight J, Percival MD, Tong V, Oballa R, Powell DA, King AJ. Characterization of CHK-336, A First-in-Class, Liver-Targeted, Small-Molecule Lactate Dehydrogenase Inhibitor for Hyperoxaluria Treatment. J Am Soc Nephrol. 2025 Apr 7;36(8):1535-1547. doi: 10.1681/ASN.0000000690. PMID 40193200